CLINICAL TRIAL: NCT03645915
Title: GLUT1: A Novel Tool Reflecting Proliferative Activity of Lung Neuroendocrine Tumors
Brief Title: GLUT1: A Novel Tool re fl Ecting Proliferative Activity of Lung Neuroendocrine Tumors
Acronym: GLUT1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0043
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Lung Tumor
Keywords: glut1; biomarkers; diagnosis
MeSH Terms: conditions — Lung Neoplasms; Disease | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunohistochemistry — Immunohistochemistry of Glut1 expression was performed in these 36 cases of neuroendocrine tumor.

SUMMARY:
Lung neuroendocrine tumor (LNT) represents approximately 20% of all lung cancers. The classification of LNT relies upon morphology. Recently, in the World Health Organization (WHO) classification, Ki-67 rate has been proposed for classi fication. It is, however, known that Ki-67 count has a poor interlaboratory reproducibly. For that reason, our team has looked for a new biomarker.

GLUT1 protein a facilitative glucose transporter protein which has ubiquitous expression in mammalian. GLUT1 is overexpressed in many human cancers. But, no study has evaluated the GLUT1 staining as an aid diagnosis in LNT.

The team have assessed the GLUT1 immunohistochemical staining in 36 LNT and to assess its diagnostic value.

DETAILED DESCRIPTION:
The (LNT) Lung neuroendocrine tumor represents approximately 20% of all lung cancers. The classification of LNT relies upon morphology. Recently, in the World Health Organization (WHO) classification, Ki-67 rate has been proposed for classi fication. It is, however, known that Ki-67 count has a poor interlaboratory reproducibly. For that reason, our team has looked for a new biomarker.

GLUT1 protein a facilitative glucose transporter protein which has ubiquitous expression in mammalian. GLUT1 is overexpressed in many human cancers. But, no study has evaluated the GLUT1 staining as an aid diagnosis in LNT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuroendocrine tumors

Exclusion Criteria:

* Patients without neuroendocrine tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between 2009 and 2014, 36 consecutive patients underwent a surgical resection or biopsy of pulmonary neuroendocrine tumor at University Hospital of Amiens: 5 cases of atypical carcinoid tumor; 13 cases of typical carcinoid tumor; 8 cases of small cell neuroendocrine carcinoma; and 10 cases of large cell neuroendocrine carcinoma. Clinical data were obtained from retrospective review of medical records: population characteristics (age, gender) and tumor size
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2016-11-13 (Actual)

PRIMARY OUTCOMES:
Assess the GLUT1 | 5years
  The objective of this study is to assess the GLUT1 staining in cohort of 36 cases of neuroendocrine tumors by immunohistochemistry and to assess its diagnostic interest.

CONTACTS AND LOCATIONS:
Overall Officials: henri sevestre, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No